CLINICAL TRIAL: NCT01622179
Title: Closed Achilles Tendon Rupture Treats by Two Different Suture Methods and the Outcome
Brief Title: Outcome of Two Different Suture Methods for Achilles Tendon Rupture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peifu Tang (Other)
Responsible Party: Sponsor-Investigator, Peifu Tang, Chief, Professor, Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PLAGH OD 13
Record Dates: First submitted 2012-06-05; First posted 2012-06-19 (Estimated); Last update posted 2013-02-20 (Estimated); Status verified 2013-02

CONDITIONS: Achilles Tendon Rupture
Keywords: surgery; suture method; blood supply

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Indirectly (Experimental): The epitenon was repaired and sewed indirectly.
  Interventions: Procedure: sewed indirectly
- Directly (Placebo Comparator): The epitenon was unrepaired and sewed directly.
  Interventions: Procedure: sewed directly

INTERVENTIONS:
Procedure: sewed indirectly — The epitenon was repaired and sewed indirectly.
  Arms: Indirectly
Procedure: sewed directly — The epitenon was unrepaired and sewed directly.
  Arms: Directly

SUMMARY:
The purpose of this study is to estimate the effective of two suture methods in the treatment of Achilles rupture.

DETAILED DESCRIPTION:
Achilles tendon rupture is one of the most common tendon injuries in the adult population. The incidence of this injury is increasing as aging adults continue their participation in high-demand sports. Although the impact of an Achilles tendon rupture is substantial, often resulting in prolonged disability and rehabilitation. Studies have showed that the operation treatment of acute Achilles tendon ruptures had some advantages. But the rebuild of blood supply was not involved in previous studies. And the epitenon of tendon is the interior layer, closest to the endotenons which contains the vascular supply. Main difference of two suture methods were if the epitenon was repaired and sewed indirectly or unrepaired and sewed directly.

ELIGIBILITY:
Inclusion Criteria:

* Adult men or women between 18 and 60 years of age.
* Closed rupture confirmed with ultrasound or magnetic resonance imaging (MRI).
* Operative within 14 days after injury.
* Willing and able to comply with and carry out the prescribed rehabilitation protocol.
* Providing informed consent.
* No other major trauma.

Exclusion Criteria:

* Refuse to participate.
* Refuse to participate.
* Additional ipsilateral injury.
* Open injury.
* Patients not suitable for surgery (i.e., mellitus diabetes, immunocompromised states, obesity (BMI.30), peripheral vascular disease or local/systemic dermatologic disorders) or have other surgical contraindications.
* Fluoroquinolone-associated rupture (i.e., rupture within 2 weeks after taking this medication).
* Achilles avulsion from the calcaneus or with bone fracture.
* Neurological or vascular disease requiring medications recognized to impair tendon healing.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-06; Primary Completion 2013-05 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Blood supply condition | six weeks
  Blood supply was estimated by ultrasonic contrast at six weeks after surgery.

SECONDARY OUTCOMES:
Calf circumference | six weeks
  Calf circumference was measured at six weeks after surgery.
Complications | six months
  Infection and rerupture at six month after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Tang P Fu, Study Chair — Chinese PLA General Hospital
Locations (1):
- Orthopedics department; The General Hospital of the People's Liberation Army, Beijing, Beijing Municipality, China